CLINICAL TRIAL: NCT03694509
Title: Gastric Emptying of Tea With Milk in Pregnancy - An Ultrasound Assessment.
Brief Title: Gastric Emptying After Tea With Milk in Pregnancy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coombe Women and Infants University Hospital (Other)
Responsible Party: Principal Investigator, Ruairi Irwin, Principal investigator, Coombe Women and Infants University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CWIUH-GUS
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Gastric Emptying
Keywords: Gastric emptying; tea; milk; pregnancy; gastric ultrasound; ultrasound; gastric antrum
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: Two groups - Tea with milk group and water control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The ultrasound assessor will be blinded to group allocation. The statistician will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breakfast tea with full fat milk (Experimental): Black breakfast tea (200ml) with full fat milk (50ml) - The volume of milk added to the tea is at the discretion of the patient but the remaining milk must be consumed afterwards.
  Interventions: Other: Breakfast tea with full fat milk
- Water (Active Comparator): Water 250ml
  Interventions: Other: Water

INTERVENTIONS:
Other: Breakfast tea with full fat milk — Assessment of gastric emptying using ultrasound. Black breakfast tea (200ml) with full fat milk (50ml) - The volume of milk added to the tea is at the discretion of the patient but the remaining milk must be consumed afterwards.
  Arms: Breakfast tea with full fat milk
Other: Water — Water 250ml.
  Arms: Water

SUMMARY:
The aim of the study is to assess the difference in gastric emptying using ultrasound of pregnant patients following a cup of tea with milk or a similar volume of water.

DETAILED DESCRIPTION:
The study involves the allocation of either 250ml of water or 200ml of tea and 50ml of milk to fasted parturients, and assessment of gastric antrum CSA at intervals up to 2 hours. The study will be performed in patients with >34 weeks gestation at the antenatal clinic. The participants will be randomized into one of two groups with an internet based randomisation tool, and then allocated to either group as per the allocation in a sealed opaque envelope. The ultrasound assessor will be blinded to the group allocation.

Participants will be asked to come to clinic in the morning fasting from solids for >6 hours and for 2 hours for clear fluids. Gastric ultrasound will be performed on the fasted pregnant patients in the right lateral decubitus position to establish a baseline and ensure that the gastric antrum is empty. Gastric antrum CSA will be measured.

Intervention group:

The intervention group will be given 200ml of black breakfast tea with 50ml of full fat milk. This should be consumed within 5 minutes. Gastric ultrasound will be performed at intervals up to 2 hours after the intervention in the right lateral decubitus position. Gastric antrum CSA will be measured. Three measurements of CSA will be taken and averaged.

Placebo group:

The placebo group will be given 250ml of water. This should be consumed within 5 minutes. Gastric ultrasound will be performed at intervals up to 2 hours after the intervention in the right lateral decubitus position. Gastric antrum CSA will be measured. Three measurements of CSA will be taken and averaged.

ELIGIBILITY:
Inclusion Criteria:

* Women with a singleton pregnancy >36 weeks.
* Subjects must be female, aged 18 years or above at baseline.
* Subjects must be able and willing to give written informed consent and to comply with the requirements of this study protocol.

Exclusion Criteria:

* Allergy/sensitivity to milk/tea.
* A medical or surgical condition leading to delayed gastric emptying (e.g. Diabetes Mellitus).
* Not fasting for 6 hours for food or 2 hours for clear fluids.
* No baseline ultrasound assessment.
* Inability to visualize the gastric antrum.
* Vomiting or inability to finish drink.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Gastric emptying at 2 hours - supine. | 120 mins
  The difference in gastric antrum cross sectional area (CSA) between groups, measured using ultrasound in a 45° semirecumbent supine position.

SECONDARY OUTCOMES:
Gastric antrum CSA - supine. | 15 mins, 30 mins, 45 mins, 60 mins, 90 mins
  The difference in gastric antrum cross sectional area (CSA) between groups, measured using ultrasound in a 45° semirecumbent supine position.
Gastric volume - supine. | 15 mins, 30 mins, 45 mins, 60 mins, 90 mins, 120 mins
  The difference in gastric volume as calculated using the determined CSA in the 45° semirecumbent supine position.
Gastric antrum CSA - RLD. | 15 mins, 30 mins, 45 mins, 60 mins, 90 mins, 120 mins
  The difference in gastric antrum cross sectional area (CSA) between groups, measured using ultrasound in the 45° semirecumbent RLD (Right lateral decubitus) position.
Gastric volume - RLD. | 15 mins, 30 mins, 45 mins, 60 mins, 90 mins, 120 mins
  The difference in gastric volume as calculated using the determined CSA in the 45° semirecumbent RLD position.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Tan, Study Director — Head of Department of Anaesthesia CWIUH
Locations (1):
- Coombe Women and Infants University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Irwin R, Gyawali I, Kennedy B, Garry N, Milne S, Tan T. An ultrasound assessment of gastric emptying following tea with milk in pregnancy: A randomised controlled trial. Eur J Anaesthesiol. 2020 Apr;37(4):303-308. doi: 10.1097/EJA.0000000000001129. PMID 31789899